CLINICAL TRIAL: NCT06373120
Title: Interventional Ventricular Assist System for PCI in Complicated and High-risk Patient: a Prospective, Multicenter, Randomized Trial
Brief Title: Interventional Ventricular Assist System for PCI in CHIP Patients
Acronym: REC-CHIPMCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QX20231057-X-1
Record Dates: First submitted 2024-03-11; First posted 2024-04-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: High-Risk Percutaneous Coronary Intervention (High-risk PCI); Left Ventricular Assist Devices
Keywords: Microaxial flow pump; ECMO; Percutaneous Coronary Intervention; left ventricular assist devices

STUDY DESIGN:
Intervention Model Description: Prospective, 1:1 randomized, controlled, multicenter trial to assess effectiveness and safety of CorVad compared to VA-ECMO in complicated and high-risk patient with indications for PCI
Who Masked: Outcomes Assessor
Masking Description: A blinded and independent clinical event adjudication committee will adjudicate all primary and secondary outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microaxial flow pump (Experimental): The microaxial flow pump (The CorVad percutaneous ventricular assist system) will offer intraoperative hemodynamic support during high-risk PCI procedures.
  Interventions: Device: Microaxial flow pump
- VA-ECMO (Active Comparator): The VA-ECMO offers intraoperative hemodynamic support during high-risk PCI procedures.
  Interventions: Device: VA-ECMO

INTERVENTIONS:
Device: Microaxial flow pump — The microaxial flow pump (The CorVad percutaneous ventricular assist system device) is a microaxial rotary blood pump that expels blood from the left ventricle into the ascending aorta, thus unloading the left ventricle. The CorVad system device can be introduced through a femoral percutaneous approach (14Fr) and can deliver an output of up to 4-6 L/min.
  Arms: Microaxial flow pump
Device: VA-ECMO — Veno-arterial extracorporeal Membrane Oxygenation (VA-ECMO) is a device originally created to replace heart and lung function. Venous deoxygenated blood is mechanically suctioned from a large central vein through a venous cannula by a centrifugal pump. It is then oxygenated, warmed, and restored into systemic circulation through an arterial cannula.
  Arms: VA-ECMO

SUMMARY:
In patients with complex coronary artery disease (CAD), determining the optimal revascularization strategy (percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) remains a challenge. These high-risk patients pose an extreme surgical risk. However, with the development of new interventional techniques and materials, PCI is a good alternative to CABG and is referred to as complex high-risk indicated PCI (CHIP).

During CHIP, hemodynamics can deteriorate because of temporary complete coronary occlusion or profound myocardial ischemia. This could result in loss of cardiac output and hemodynamics collapse. Mechanical support during CHIP facilitates native cardiac function by achieving a stable hemodynamic state to withstand repetitive derangements such as ischemia caused by prolonged and repeated balloon inflations, and resume original cardiac function immediately postprocedure or shortly thereafter.

There are several mechanical circulatory support (MCS) systems available, i.e., intra-aortic balloon counterpulsation (IABP), Impella, TandemHeart, and veno-arterial extracorporeal membrane oxygenation (VA-ECMO). These MCS have been widely studied in patients with acute myocardial infarction (MI) complicated by cardiogenic shock and showed conflicting results. However, studies regarding the use of MCS in the setting of CHIP are much less abundant and no randomized study has compared Impella with VA-ECMO in CHIP patients.

The aim of the study is to evaluate the effectiveness of interventional ventricular assist system (CorVad) compared to the venoarterial extracorporeal membrane oxygenation (VA-ECMO) system in providing circulatory support for complicated and high-risk patient with indications for PCI.

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years to 90 Years
2. The Heart Team determined that the patients required coronary artery revascularization, but there is a high risk of CABG or the patients refuses CABG. After evaluation by the Heart Team, it was concluded that the patients can benefit from revascularization by undergoing high risk PCI
3. The subject is diagnosed with acute or chronic coronary syndrome, and

   1. LVEF≤ 35% or
   2. LVEF ≤ 40% and NYHA Classification is III or IV
4. Patients who are able to give informed consent and complete the follow-up

Image inclusion criteria

1. At least two vessel chronic total occlusions (CTOs) (diameter of occluded artery ≥ 2.5mm)
2. Unprotected left main coronary artery disease, and meeting one or more complex PCI maneuver criteria
3. Three-vessel disease and meeting two or more complex PCI criteria

Complex PCI maneuvers are defined as:

1. Bifurcation require the treatment of both branches (including stents or PTCA)
2. Calcification require Excimer laser coronary atherectomy, intravascular lithotripsy, or rotational atherectomy
3. Severe tortuosity
4. Target lesion is CTO (diameter of occluded artery ≥ 2.5mm and J-CTO score ≥ 2 points)

Exclusion Criteria

1. Had mechanical circulatory support treatment (such as IABP, ECMO, pVAD) before randomization
2. Acute myocardial infarction or with thrombolytic treatment within 7 days
3. Cardiopulmonary resuscitation within 24 hours
4. Cardiogenic shock (systolic blood pressure < 90 mmHg for more than 30 minutes or requiring vasoactive drugs to maintain systolic blood pressure above 90 mmHg) or hemodynamically unstable
5. pVAD and ECMO cannot be inserted or contraindicated (including but not limited to left ventricular mural thrombus, artificial aortic valve or cardiac contraction device, moderate to severe aortic stenosis, moderate to severe aortic valve insufficiency, peripheral stents, tortuosity, dissection and other severe vascular diseases obstructing the insertion of the study device, aortic dissection, aneurysm or severe abnormalities of the ascending aorta and/or aortic arch, red blood cell fragility or blood disorders, hypertrophic obstructive cardiomyopathy)
6. Abnormal coagulation function (routine blood test indicates platelet count less than 50×109/L, or more than 700×109/L)
7. Active visceral bleeding occurred within 1 month
8. Ischemic or hemorrhagic stroke occurred within 1 month
9. Known contraindication to antiplatelet and anticoagulant medications
10. Known contraindication to medications such as Heparin or contrast.
11. Need for dialysis treatment
12. Active infection
13. Expected life span of less than one year
14. Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential according to local practice)
15. Currently participating in another trial and not yet at its primary endpoint
16. Severe pulmonary arterial hypertension
17. Severe right heart failure or severe tricuspid regurgitation
18. Unforeseen circumstances that the researcher has deemed to be inappropriate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Major adverse event | 1 month
  Major adverse event is a composite endpoint, defined as all-cause death, stroke, myocardial infarction, revascularization, cardiovascular hospitalization, MCS-ARC defined bleeding types 3, 4, or 5, acute kidney injury, serious device-related adverse events, cardiopulmonary resuscitation

SECONDARY OUTCOMES:
All-cause death | 1, 3, 12, 24, 36, and 60 months
Stroke | 1, 3, 12, 24, 36, and 60 months
Myocardial infarction | 1, 3, 12, 24, 36, and 60 months
Revascularization | 1, 3, 12, 24, 36, and 60 months
Cardiovascular hospitalization | 1, 3, 12, 24, 36, and 60 months
  Rehospitalization due to cardiovascular reasons
MCS-ARC defined type 3, 4, 5 bleeding | 1 month
  Bleeding is defined by the "Updated deﬁnitions of adverse events for trials and registries of mechanical circulatory support: A consensus statement of the mechanical circulatory support academic research consortium" (MRC-ARC)
Acute kidney injury | 1 month
Serious device-related adverse events | 1 month
  Including but not limited to cardiac structural impairment, severe limb ischemia (pale, pulseless, and necrotic), infection, aortic and aortic valve impairment, hemolysis, peri-procedural complications that cause death, permanent/severe disability to the subject, or significantly prolonged hospital stay or need for surgical intervention
Cardiopulmonary resuscitation | 1 month
Hospitalization time | 1 month
Intensive care unit (ICU/CCU) stay time | 1 month
ECMO/Corvad utilization time | 1 month
Hemodynamic disorder | 1 month
  Hemodynamic disorder is defined as average arterial pressure (MAP) below 60 mmHg for more than 10 minutes with the requirement of additional vasoactive medications
Transfusion rate | 1 month
  Transfusion rate is defined as patients who had transfusion / all enrolled patients.
Units of transfusion | 1 month
Major adverse event | 3, 12, 24, 36, and 60 months
  Major adverse event is a composite endpoint, defined as all-cause death, stroke, myocardial infarction, revascularization, cardiovascular hospitalization, MCS-ARC defined bleeding types 3, 4, or 5, acute kidney injury, serious device-related adverse events, cardiopulmonary resuscitation
Major Adverse Cardiovascular and Cerebrovascular Events | 1, 3, 12, 24, 36, and 60 months
  Major Adverse Cardiovascular and Cerebrovascular Events is a composite endpoint, defined as all-cause death, stroke, myocardial infarction, revascularization, cardiovascular hospitalization

OTHER OUTCOMES:
Device-related composite endpoint (DoCE) | 1, 3, 12, 24, 36, and 60 months
  Device-related composite endpoint (DoCE), defined as: cardiac death, target-vessel myocardial infarction (TV-MI), clinically and physiologically driven target lesion revascularization (CPI-TLR)
Patient-related composite endpoint (PoCE) | 1, 3, 12, 24, 36, and 60 months
  Patient-related composite endpoint (PoCE), defined as: all-cause death, any stroke, any myocardial infarction, and any revascularization
Net adverse clinical events | 1, 3, 12, 24, 36, and 60 months
  Net adverse clinical events, defined as: PoCE + MCS-ARC defined type 3, 4, 5 bleeding
Cardiac death | 1, 3, 12, 24, 36, and 60 months
Ischemic stroke | 1, 3, 12, 24, 36, and 60 months
Hemorrhagic stroke | 1, 3, 12, 24, 36, and 60 months
Transient ischemic attack | 1, 3, 12, 24, 36, and 60 months
Target vessel myocardial infarction | 1, 3, 12, 24, 36, and 60 months
Target lesion revascularization | 1, 3, 12, 24, 36, and 60 months
Target vessel revascularization | 1, 3, 12, 24, 36, and 60 months
Clinically and physiologically driven target lesion revascularization (CPI-TLR) | 1, 3, 12, 24, 36, and 60 months
Rehospitalization | 1, 3, 12, 24, 36, and 60 months
MCS-ARC type 2 bleeding | 1 month
Puncture complications | 1 month
  Puncture complications: Vascular complications or percutaneous vascular suture failure
Aortic valve injury | 1 month
  Aortic valve injury is defined as the occurrence of moderate and severe aortic valve regurgitation in patients with no pre-operative aortic valve regurgitation or mild regurgitation
Active Infection | 1 month
  Active infection refers to an infection accompanied by clinical evidence, including pain, fever, or imaging findings consistent with infection, and requires the use of antimicrobial drugs for treatment. The definition of infection requires positive culture results from the site or organ of infection, unless there is strong clinical evidence indicating the presence of infection and the need for treatment.
ECMO/Corvad setup time | assessed at index PCI procedure
  Setup time is defined as the time from starting vessel puncture to the time providing cardiac support by the device
Complete revascularization rate | 1 month
  Complete revascularization is defined as the residual SYNTAX score ≤ 8 points
Change in left ventricular ejection fraction (LVEF) from baseline | 1, 12, 24, 36, and 60 months
Change in New York Heart Association (NYHA) classification from baseline | 1, 12, 24, 36, and 60 months
Change in Seattle Angina Questionnaire (SAQ) score from baseline | 1, 12, 36, and 60 months
  The SAQ is a 19-item self-administered disease-specific patient-reported outcome measure with 5 domains: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception and/or quality of life. It was to identify a conceptual framework with which to elicit the important manifestations of coronary disease from the patient perspective. All SAQ domain scores and the summary score range from 0 to 100 points, with higher scores indicating less angina, fewer functional limitations, and better quality of life.
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score from baseline | 1, 12, 36, and 60 months
  The KCCQ is a self-administered, 23-item questionnaire that quantifies physical limitations, symptoms, self-efficacy, social interference and quality of life. KCCQ scores range from 0 to 100, with higher scores indicating fewer symptoms and physical limitations.
Change in 5-level EQ-5D version (EQ-5D-5L) standardized health status scale score from baseline | 1, 12, 36, and 60 months
  The EQ-5D is a standardized instrument for use as a measure of health outcome which can be divided into two parts: the EQ-5D health description system and the EQ-vas. EQ-5D-5L questionnaire is a five-item scale assessing five separate dimensions of health: (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has to be answered on a five-level scale (no problems, slight problems, moderate problems, severe problems and extreme problems). The EQ-VAS is a 20 cm long vertical visual scale. A score of 100 at the top represents "best perceived health status" and a score of 0 at the bottom represents "worst perceived health status".
Change in creatinine clearance rate from baseline | 1 month
Stent thrombosis | 1, 3, 12, 24, 36, and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D., Study Chair — Xijing Hospital; Chao Gao, M.D., Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China